CLINICAL TRIAL: NCT03314493
Title: Effect of Spironolactone on the Progression of Coronary Calcification in Peritoneal Dialysis Patients
Brief Title: Prevention of the Progression of Coronary Calcification With Use of Spironolactone in Peritoneal Dialysis Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Professor Fernando Figueira Integral Medicine Institute (Other)
Collaborators: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Alex Sandro Rolland de Souza, Professor, Professor Fernando Figueira Integral Medicine Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: U1111-1203-1767
Record Dates: First submitted 2017-10-04; First posted 2017-10-19 (Actual); Last update posted 2017-10-19 (Actual); Status verified 2017-10

CONDITIONS: Coronary Artery Calcification; Vascular Calcification
Keywords: Vascular calcification; Coronary calcification; Peritoneal Dialysis; Spironolactone
MeSH Terms: conditions — Vascular Calcification | interventions — Spironolactone; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | US Export: No

ARMS (2):
- Spironolactone group (Experimental): Spironolactone oral tablet 25mg/day, for 12 months
  Interventions: Drug: Spironolactone 25Mg Tablet
- Control group (No Intervention): No spironolactone use

INTERVENTIONS:
Drug: Spironolactone 25Mg Tablet — Patients with coronary calcium score > 30 were treated with spironolactone for 12 months
  Arms: Spironolactone group

SUMMARY:
Vascular calcification is a frequent complication in dialysis patients and is strongly associated with mortality. Its pathogenesis is complex and involves a series of markers that act on the vascular microenvironment. There is evidence that aldosterone is one of the biomarkers and may have a role in osteoinductive pathways.The aim of this study was to evaluate the effect of spironolactone, an inhibitor of mineralocorticoid receptor, in the progression of coronary calcification in patients undergoing peritoneal dialysis.

ELIGIBILITY:
Inclusion Criteria:

* Coronary calcium score > 30 Agatston unit
* Peritoneal dialysis for at least 6 months

Exclusion Criteria:

* Use of spironolactone in the last 3 months
* Mean serum potassium > 6 mEq/L in the last 3 months
* Cardiac revascularization surgeries
* Arrhythmias
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2014-11-07 (Actual); Primary Completion 2016-11-10 (Actual); Study Completion 2016-11-10 (Actual)

PRIMARY OUTCOMES:
Relative progression of the coronary calcium score | 12 months
  Percentage change in coronary calcium score from baseline to end of study. Coronary calcium score detected using multi-detector computed tomography and expressed in Agatston units.

SECONDARY OUTCOMES:
Absolute progression of the coronary calcium score | 12 months
  To evaluate the absolute progression of the coronary calcium score, defined as the difference between the final score and the baseline score. Coronary calcium score detected using multi-detector computed tomography and expressed in Agatston units.
Adverse effects of spironolactone use | 12 months
  During follow-up, all patients were assessed monthly to evaluate the frequency of hyperpotassemia (serum potassium > 6mEq/L), hypotension (systolic blood pressure < 100 mmHg) and/or diastolic blood pressure < 60 mmHg) and gynecomastia defined as breast augmentation, painful or not.
1 year change in laboratory parameters of mineral metabolism | 12 months
  Assess changes in serum levels of total calcium, phosphorus, alkaline phosphatase, 25(OH) vitamina D and intact parathyroid hormone, through periodic blood dosages of these parameters, during follow-up.
Need for spironolactone dose reduction | 12 months
  In the presence of adverse effects, the dose of spironolactone was reduced from 25 to 12,5 mg per day.
Causes of discontinuation of the study | 12 months
  Severe hyperpotassemia defined as serum potassium>7mEq/L; lack of improvement in the adverse effects of spironolactone with a dose reduction of 12,5 mg/day, ie, persistence of breasts enlargement, hypotension and hyperpotassemia (serum potassium < 6mEq/L); discontinuation of peritoneal dialysis due to renal transplantation or the need for hemodialysis transfer; withdrawal of consent at any time; and death were considered as causes for discontinuation of the study. For the evaluation of this outcome, the patients were submitted to medical visit and biochemical measures monthly.
1 year change in laboratory parameters related to inflammation. | 12 months
  Assess changes on serum levels of c-reactive protein, albumin and fetuin-A, through periodic blood dosages of these parameters, during follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Paula S Gueiros, MD, Principal Investigator — Instituto de Medicina Integral Prof. Fernando Figueira; Alex SR Souza, PhD, Principal Investigator — Instituto de Medicina Integral Prof. Fernando Figueira; Aluizio B Carvalho, PhD, Study Director — Universidade Federal de São Paulo; José E Gueiros, MD, Study Chair — Instituto de Medicina Integral Prof. Fernando Figueira; Leuridan T Cavalcante, PhD, Study Chair — Instituto de Medicina Integral Prof. Fernando Figueira; Dulce E Casarini, PhD, Study Chair — Universidade Federal de São Paulo; Marina M Cadena, Study Chair — Instituto de Medicina Integral Prof. Fernando Figueira; Karina T Nobrega, MD, Study Chair — Instituto de Medicina Integral Prof. Fernando Figueira; Eveline B Calado, MD, Study Chair — Instituto de Medicina Integral Prof. Fernando Figueira
Locations (1):
- Instituto de Medicina Integral Prof. Fernando Figueira, Recife, Pernambuco, Brazil

REFERENCES:
- [Background] Fischer SS, Kempe DS, Leibrock CB, Rexhepaj R, Siraskar B, Boini KM, Ackermann TF, Foller M, Hocher B, Rosenblatt KP, Kuro-O M, Lang F. Hyperaldosteronism in Klotho-deficient mice. Am J Physiol Renal Physiol. 2010 Nov;299(5):F1171-7. doi: 10.1152/ajprenal.00233.2010. Epub 2010 Aug 18. PMID 20719979
- [Background] Voelkl J, Alesutan I, Leibrock CB, Quintanilla-Martinez L, Kuhn V, Feger M, Mia S, Ahmed MS, Rosenblatt KP, Kuro-O M, Lang F. Spironolactone ameliorates PIT1-dependent vascular osteoinduction in klotho-hypomorphic mice. J Clin Invest. 2013 Feb;123(2):812-22. doi: 10.1172/JCI64093. Epub 2013 Jan 9. PMID 23298834
- [Background] Tatsumoto N, Yamada S, Tokumoto M, Eriguchi M, Noguchi H, Torisu K, Tsuruya K, Kitazono T. Spironolactone ameliorates arterial medial calcification in uremic rats: the role of mineralocorticoid receptor signaling in vascular calcification. Am J Physiol Renal Physiol. 2015 Dec 1;309(11):F967-79. doi: 10.1152/ajprenal.00669.2014. Epub 2015 Sep 2. PMID 26336165
- [Result] Nitta K, Akiba T, Nihei H. Aldosterone blockade and vascular calcification in hemodialysis patients. Am J Med. 2003 Aug 15;115(3):250. doi: 10.1016/s0002-9343(03)00293-6. No abstract available. PMID 12935835
- [Result] Matsumoto Y, Mori Y, Kageyama S, Arihara K, Sugiyama T, Ohmura H, Yakushigawa T, Sugiyama H, Shimada Y, Nojima Y, Shio N. Spironolactone reduces cardiovascular and cerebrovascular morbidity and mortality in hemodialysis patients. J Am Coll Cardiol. 2014 Feb 18;63(6):528-36. doi: 10.1016/j.jacc.2013.09.056. Epub 2013 Oct 30. PMID 24184249
- [Derived] Hasegawa T, Nishiwaki H, Ota E, Levack WM, Noma H. Aldosterone antagonists for people with chronic kidney disease requiring dialysis. Cochrane Database Syst Rev. 2021 Feb 15;2(2):CD013109. doi: 10.1002/14651858.CD013109.pub2. PMID 33586138